CLINICAL TRIAL: NCT02757976
Title: Resynchronization for Ambulatory Heart Failure Trial - LV Endocardial
Acronym: RAFT-LVendo
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Consensus RAFT-LVendo Steering Committee to terminate.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 252410
Record Dates: First submitted 2016-04-28; First posted 2016-05-02 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Heart Failure, Left Ventricular Dysfunction
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Left

STUDY DESIGN:
Intervention Model Description: This trial will compare two management strategies for patients with Heart Failure, left ventricular systolic dysfunction, and intermediate prolonged QRS duration (120-149ms). The control group is conventional Cardiac Resynchronization Therapy (CRT). The experimental group is LV endocardial CRT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional CRT (Active Comparator): Patients randomized to the Conventional CRT will receive a CRT device with or without ICD. Device implantation will be performed within 10 working days of randomization. Conscious sedation or general anesthesia can be used for the implant procedure. The device will be implanted in a facility that has the capacity to perform coronary sinus venography at the time of implantation. The RA lead will be placed in the RA appendage or high RA. The RV lead should be placed at the RV apex or distal RV septum (R wave > 7 mV, pacing threshold < 1.5 V at a pulse-width of 0.5 ms). The LV lead should be positioned through the CS to an LV branch. The lead should be placed at one of the left ventricular venous branches, avoiding the LV apex and scar region identified by pre-implant imaging
  Interventions: Device: Conventional CRT
- LV endocardial CRT (Experimental): Patients randomized to LV endocardial CRT will receive a CRT device with or without ICD, placed in the same time frame, and will have RA and RV leads implanted as the conventional CRT group. The device will be implanted in a facility that has the capacity to perform trans-atrial septal puncture with ultrasound guidance (TEE or ICE) at the time of implantation. The LV lead will be placed using a trans-atrial septal approach, using a specially designed puncture tools and LVendo delivery tool kits specifically designed for this study. Special care will be taken to avoid the LV apex and transmural scar identified by pre-implant imaging.
  Interventions: Device: LV endocardial CRT

INTERVENTIONS:
Device: Conventional CRT — Patients randomized to the Conventional CRT will receive a CRT device with or without ICD. Device implantation will be performed within 10 working days of randomization. Conscious sedation or general anesthesia can be used for the implant procedure. The device will be implanted in a facility that has the capacity to perform coronary sinus venography at the time of implantation. The RA lead will be placed in the RA appendage or high RA. The RV lead should be placed at the RV apex or distal RV septum (R wave > 7 mV, pacing threshold < 1.5 V at a pulse-width of 0.5 ms). The LV lead should be positioned through the CS to an LV branch. The lead should be placed at one of the left ventricular venous branches, avoiding the LV apex and scar region identified by pre-implant imaging.
  Arms: Conventional CRT
Device: LV endocardial CRT — Patients randomized to LV endocardial CRT will receive a CRT device with or without ICD, placed in the same time frame, and will have RA and RV leads implanted as the conventional CRT group. The device will be implanted in a facility that has the capacity to perform trans-atrial septal puncture with ultrasound guidance (TEE or ICE) at the time of implantation. The LV lead will be placed using a trans-atrial septal approach, using a specially designed puncture tools and LVendo delivery tool kits specifically designed for this study. Special care will be taken to avoid the LV apex and transmural scar identified by pre-implant imaging.
  Arms: LV endocardial CRT

SUMMARY:
This trial will compare two strategies for patients with Heart Failure, Left Ventricular systolic dysfunction, and intermediate QRS durations. The control group is conventional CRT. The experimental group is LVendo CRT

DETAILED DESCRIPTION:
Patients randomized to the Conventional CRT will receive a CRT device with or without ICD. Device implantation will be performed within 10 working days of randomization.

Patients randomized to LV endocardial CRT will receive a CRT device with or without ICD, placed in the same time frame and will have RA and RV leads implanted as the conventional CRT group. The device will be implanted in a facility that has the capacity to perform trans-atrial septal puncture with ultrasound guidance. The LV lead will be placed using a trans-atrial septal approach using a specially designed puncture tools and LVendo delivery tool kits specifically designed for this study

ELIGIBILITY:
Inclusion Criteria:

* Patients with NYHA Class II or III or ambulatory IV HF symptoms
* Optimal HF Medical Therapy of at least 3 months (2009 ACCF/AHA, ESC 2012)
* LVEF less than or equal to 35%
* Sinus rhythm (can have paroxysmal atrial fibrillation)
* QRS morphology is non-RBBB
* QRS durations more than or equal to 120 ms, but less than 150 ms
* Patients are able to receive chronic oral anticoagulation
* Patients with pacemaker or ICD that meet the above criteria may be upgraded to CRT-D or CRT-P

Exclusion Criteria:

* Planned Atrial Fibrillation Ablation within 12 months
* Patients with mitral or tricuspid prosthetic valve that precludes the placement of an LV lead transvenously or trans-septally
* Patients with RBBB
* Patients with LV thrombus
* Patients with permanent atrial fibrillation
* Patients with contraindications to oral anti-coagulation
* In-hospital patients with acute cardiac or non-cardiac illness that requires intensive care
* Acute coronary syndrome (including MI) < 4 weeks
* Coronary revascularization (CABG or PCI) < 3 months
* Uncorrected or uncorrectable primary valvular disease
* Restrictive, hypertrophic or reversible form of cardiomyopathy
* Severe primary pulmonary disease such as cor pulmonale
* Expected to undergo cardiac transplantation within one year (status I)
* Patients with a life expectancy of less than one year from non-cardiac cause.
* Patients included in other clinical trials that will affect the objectives of this study
* Those unable or unwilling to provide informed consent
* Those with a history of noncompliance to medical therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Assessment of LVESVi | Baseline to 6 months & 12 months
  LV reverse remodeling as measured by the difference of LVESVi on echocardiography (echo)

SECONDARY OUTCOMES:
Ventricular arrhythmia burden determined by the device capture of arrhythmias and adjudication by a device review committee blinded to patient's treatment allocation. | Baseline to 6 months & 12 months
NT-proBNP measurement | Baseline to 6 months & 12 months
6 Minute Hall Walk Distance | Baseline to 6 months & 12 months
Quality of Life Measure | Baseline to 6 months & 12 months
  EQ5D-5L & Minnesota Living with HF
Mortality | Baseline to 6 months & 12 months
Heart Failure Admissions | Baseline to 6 months & 12 months
Reduction of LVEF | Baseline to 6 months & 12 months

OTHER OUTCOMES:
Thromboembolic Events Investigator deemed to be directly related to the therapy | Baseline to 12 months
  Safety
Safety: LVendo CRT: specific system placement procedure related adverse events | Baseline to 12 months
  Safety
Safety:Pocket infection requiring extending hospitalization > 24 hours or requiring surgical intervention | Baseline to 12 months
Safety:Lead(s) dislodgement requiring repositioning or cessation of CRT | Baseline to 12 months
Safety:Cardiac tamponade requiring intervention | Baseline to 12 months
Safety:Phrenic nerve stimulation | Baseline to 12 months

CONTACTS AND LOCATIONS:
Locations (11):
- Canada (11):
  - Libin Cardiovascular Institute, Calgary, Alberta
  - Royal Columbia Hospital, New Westminster, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Queen Elizabeth II Health Science, Halifax, Nova Scotia
  - London Health Science Centre, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael Hospital, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Institut Univ.cardiologie/pneumologie de Québec, Québec, Quebec
  - CHUS Le Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No